CLINICAL TRIAL: NCT01595542
Title: A School Health Center Intervention to Increase Adolescent Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-1041
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Immunization Program; School Health Services; HPV Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Parents served by experimental school sites received intervention packets including modified vaccine consent form
  Interventions: Behavioral: Modified Vaccine Consent Form
- Control (No Intervention): Did not receive intervention materials

INTERVENTIONS:
Behavioral: Modified Vaccine Consent Form — Packet of written immunization materials for parents and students which includes the following:
  1. Cover letter
  2. Vaccine promotional flyer
  3. Vaccine information sheets (one for adolescent vaccination and one for other vaccination)
  4. Improved consent form
  5. Note advertising a lottery for free movie tickets for returning the consent form
  6. Self-addressed stamped envelope
  Arms: Intervention

SUMMARY:
The study will evaluate a health services intervention to increase uptake of adolescent vaccines (HPV, Tdap, meningococcal conjugate, and influenza) among students enrolled in five school health centers by improving the consent process for parents.

ELIGIBILITY:
Inclusion Criteria:

* All students enrolled at target schools

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3417 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change from Baseline In The Number of Adolescent Vaccines | 4 months post intervention
  Change in vaccination rates for HPV, Tdap, meningococcal conjugate and influenza between Fall 2011 (baseline) and Fall 2012.

SECONDARY OUTCOMES:
Number of Returned Consent Forms Authorizing Vaccination | 4 months post intervention
  Number of signed and returned consent forms for adolescent vaccines HPV, Tdap, meningococcal conjugate and influenza in the intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Noel T Brewer, PhD, Principal Investigator — University of North Carolina Chapel Hill, Department of Health Behavior and Health Education
Locations (1):
- Student Health Centers, Chapel Hill, North Carolina, United States